CLINICAL TRIAL: NCT01051310
Title: Feasibility Study of Percutaneous Aortic Valve Implantation With the Medtronic CoreValve System for Percutaneous Aortic Valve Replacement (PAVR) in Patients With a Failing Previously Surgically Implanted Aortic Bioprosthesis and Presenting a High Risk for Repeat Surgical Valve Replacement
Brief Title: Medtronic CoreValve REDO Study
Acronym: REDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COR-2007-03
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CoreValve (Experimental)
  Interventions: Device: Medtronic CoreValve System

INTERVENTIONS:
Device: Medtronic CoreValve System — Transcatheter Aortic Valve
  Other Names: Medtronic CoreValve Transcatheter aortic valve; Medtronic CoreValve Percutaneous aortic valve

SUMMARY:
The proposed investigation is a prospective, multicenter, non-randomized study to evaluate the immediate benefits (at discharge and at 30 days) in terms of performance and safety of the implantation of the Medtronic CoreValve PAV in a failing aortic bioprosthesis. In addition, the study aims to evaluate the performance and the safety of the implantation of the Medtronic CoreValve PAV in a failing aortic bioprosthesis at subsequent annual follow-ups out to 48 months post procedure.

These objectives will be achieved through the following endpoints:

* Primary safety endpoint - Composite of Major Adverse Events
* Primary performance endpoint - Technical and procedural success at discharge

Patient Population: Eligible subjects will be at least 75 years old, presenting with a failing aortic bioprosthesis (stenotic, incompetent or mixed) including homograft or stented or stentless heterograft, considered poor surgical candidates and necessitating repeat aortic valve replacement. Up to 20 patients will be included in up to four hospitals.

ELIGIBILITY:
Inclusion Criteria:

* > 74 years old,
* Symptomatic failing bioprosthetic aortic valve (stenotic, incompetent or mixed) confirmed by Doppler echocardiography,
* Logistic EuroSCORE > 15%, or
* Any of the following criteria:

  1. Left ventricular ejection fraction (LVEF) < 20%,
  2. Creatinine clearance < 20mL/min (estimation using the Cockcroft calculation),
  3. Renal failure requiring dialysis,
  4. Permanent and long lasting (> 6 month duration) atrial fibrillation,
  5. Cirrhosis of the liver (Child class A or B),
  6. Respiratory impairment (FEV1 < 1L),
  7. Previous cardiac surgery (i.e., CABG especially if patient had competent mammary arteries on left anterior descending (LAD) artery or occluded saphenous veins with high-risk of coronary embolism during re-operation),
  8. Pulmonary hypertension ³ 60mmHg,
  9. Recurrent pulmonary embolus,
  10. Moderate tricuspid (< grade 2+) insufficiency,
  11. Any severe disease contraindicating surgery,
  12. Calcified aorta (porcelain aorta),
  13. Recent myocardial infarction (less than 30 days at baseline),
  14. Contraindication for cardiopulmonary bypass,
* Inner diameter of the failing bioprosthetic aortic valve (homograft or stented or stentless heterograft) of ³ 19mm and < 26mm as determined by Doppler echocardiography,
* Signed informed consent form.

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine and clopidogrel, Nitinol, or sensitivity to contrast media which cannot be pre-medicated,
* Active infection or endocarditis,
* Any intra left ventricular mass, thrombus or vegetation evidenced by Doppler echocardiography,
* Mitral or tricuspid valvular insufficiency ³ grade 2+,
* Prosthetic mitral or tricuspid valve,
* Femoral and/or iliac and/or aortic vascular condition (stenosis, occlusion or tortuosity) that could complicate endovascular access to the aortic valve bioprosthesis,
* Symptomatic carotid or vertebral artery narrowing (> 70%) disease,
* Aortic abdominal or thoracic aneurysm,
* Bleeding diathesis or coagulopathy, or patient refuses blood transfusion,
* Active peptic ulcer or has had upper gastrointestinal bleeding within the past 3 months before baseline,
* Moribund status or cachexia with short life-expectancy independent of cardiac condition,
* Any acute neurological event or dysfunction occurred in the past 6 weeks before baseline or patient with severe senile dementia,
* Therapeutic invasive cardiac procedure, other than balloon aortic valvuloplasty, performed within 30 days prior to study procedure or to be performed during or within 30 days after the study procedure,
* Currently, enrolled in this study or another investigational drug or device study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Grube, Prof. Dr., Principal Investigator — Helios Heart Center Siegburg, Germany; G. Schuler, Prof. Dr., Principal Investigator — Universitat Leipzig Herzzentrum, Germany; R. Lange, Prof. Dr., Principal Investigator — Deutsches Herzzentrum Munich, Germany; P. de Jaegere, Dr., Principal Investigator — Erasmus MC Rotterdam, Netherlands
Locations (3):
- Germany (2):
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, München
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- See also: Related Info — http://www.medtronic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three sites in Germany enrolled 18 patients between June 2008 and January 2010.
Pre-assignment Details: All 18 subjects signed and informed consent and were admitted to the catheterization laboratory for an attempted implantation. All 18 subjects were subsequently implanted with the CoreValve device.
Groups:
- Overall Study: All enrolled subjects who received the Medtronic CoreValve aortic valve prosthesis
Period: Overall Study
Arm/Group | Overall Study
Started | 18
Completed | 13
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received the Medtronic CoreValve aortic valve prosthesis
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of MAE Free Subjects
Description: Percentage of subjects without a composite major adverse event (MAE) at 30 days post procedure. the composite MAE includes:
  1. MACCE (Major Adverse Cardiac or Cerebral Event): cardiac death, documented Mobitz type II second degree and third degree atrioventricular block, neurological events and surgical aortic valve replacement.
  2. MAE: non cardiac death including sudden unexpected or unexplained death, cardiac tamponade, nonstructural valve dysfunction resulting in stenosis or regurgitation at the study valve not intrinsic to the valve itself, structural valve deterioration cardiogenic shock, operated valve endocarditis, valve thrombosis, aortic dissection/perforation, major bleeding event, peripheral embolic event and emergent revascularization procedure.
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Participants | 10

2. Primary Outcome: Technical Success.
Description: The number of subjects in whom technical success was achieved where technical success was defined based on the device functionality as judged by the investigator adressing the ability of the system (1) to access the failing bioprosthetic valve via a peripheral vessel with the delivery catheter and (2) to deploy the valve accurately across the failing bioprosthetic valve and (3) to remove intact delivery system.
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Participants | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected from implantation till 12 months follow up
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 5/18
Serious Adverse Events (participants affected / at risk) | 15/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=18)
Myocardial infarction (Cardiac disorders) | 1 (1)
Documented Mobitz type II AVB II, AVB III (Cardiac disorders) | 5 (25)
(General disorders) | 12 (19) — Any other reported adverse event not associated with the use of the study device were collected without a specific adverse event term
bleeding event (Injury, poisoning and procedural complications) | 2 (2)
Neurological events (CVA, RIND, TIA) (Nervous system disorders) | 2 (2)
non structural valve dysfunction (Product Issues) | 1 (1)
Surgical aortic valve replacement (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=18)
(General disorders) | 13 (44) — Any other reported adverse event not associated with the use of the study device were collected without a specific adverse event term
bleeding event (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No